CLINICAL TRIAL: NCT06503133
Title: The Effect of Online Prenatal Yoga-Assisted Birth Preparation Training Based on Albert Bandura's Self-Efficacy Theory on Fear of Childbirth and Childbirth Self-Efficacy in Primiparas: Randomized Controlled Study
Brief Title: The Effect of Prenatal Yoga-Assisted Birth Preparation Training on Fear of Childbirth and Childbirth Self-Efficacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Eda Simsek Sahin, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-664219
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Fear of Childbirth; Childbirth Self Efficacy
Keywords: Birth preperation training; Prenatal yoga; Fear of childbirth; Childbirth self efficacy

STUDY DESIGN:
Intervention Model Description: The research is a single-centre parallel randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant blinding is planned to prevent bias in the research. At the beginning of the study, all participants will be informed that prenatal yoga-supported online birth preparation training will be applied, but the start times of prenatal yoga practice may vary depending on the groups to which they will be randomly assigned, and they will be assigned to the experimental and control groups by randomization by an independent researcher. After the final measurements are taken, the participants in the control group will also undergo prenatal yoga practice. In addition, the independent researcher will make the post-test measurements. Data collected by the independent researcher will be ambiguously coded as A and B. The data will be analyzed and reported by an independent statistician. The groups will be unclear during the analysis and reporting phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Yoga-Supported Birth preparation Training Group (Experimental): Participants in this group will receive a 6-week prenatal yoga-supported birth preparation training program based on Albert Bandura's self-efficacy theory.
  Interventions: Other: Birth preparation training; Other: Prenatal yoga practice
- Birth Preparation Training Group (Active Comparator): Participants in this group will receive a 6-week birth preparation training program based on Albert Bandura's self-efficacy theory.
  After the post-test measurements are taken, participants in this group will also be offered the opportunity to apply prenatal yoga.
  Interventions: Other: Birth preparation training

INTERVENTIONS:
Other: Birth preparation training — Birth preparation training is based on Albert Bandura's self-efficacy theory. It is a 60-minute training once a week. The first 10 minutes of the training are devoted to the initial activity, 40 minutes to sharing the training content, and 10 minutes to answering the participants' questions and receiving feedback. The training will be conducted in closed groups via the online meeting program (Zoom®).
Other: Prenatal yoga practice — Prenatal yoga practice is a 60-minute practice once a week. The first 5 minutes of the prenatal yoga practice are devoted to guided meditation, 40 minutes to active asanas (yoga pose), 5 minutes to pranayama practice (breathing exercise) and 10 minutes to savasana (relaxing yoga pose). Prenatal yoga practice will be conducted in closed groups via the online meeting program (Zoom®)
  Arms: Prenatal Yoga-Supported Birth preparation Training Group

SUMMARY:
Pregnancy is a life event that requires biopsychosocial adaptation. Although pregnancy is often perceived as a positive and physiological process, women experience a wide range of fears of childbirth, from simple anxiety to severe phobic fear (tokophobia), during their pregnancy. It is thought that the feeling of experiencing pain often lies at the root of the fear of childbirth. However, fear of childbirth can be experienced for many different reasons depending on biological, psychological and sociocultural factors, personal characteristics and experiences. The prevalence of fear of childbirth in the world is 14%. In Turkey, the prevalence of fear of childbirth varies between 16% and 69%, and 21% of women experience fear of childbirth at a clinical level. In general, fear is a physiological reaction that is important for the safety of the individual, and it is thought that low-level fear of childbirth will prepare individuals for parenting. However, uncontrollable fear of childbirth can lead to physical, emotional and behavioural changes that negatively affect the woman's daily life, prolonged labour and childbirth complications. Most importantly, women who cannot cope with the fear of childbirth may perceive cesarean section as the only solution and turn to elective cesarean section. The total cesarean section rate in Turkey is 52%, which is much higher than the World Health Organization's acceptable cesarean section rate. Fear of childbirth has been accepted as an important public health problem that needs intervention both in the world and in our country, and research on fear of childbirth has accelerated, especially in the last twenty years.

DETAILED DESCRIPTION:
Although there are many factors affecting fear of childbirth, childbirth self-efficacy is among the important predictors of fear of childbirth. Albert Bandura defines self-efficacy as "an individual's belief in his or her ability to engage in behaviour that leads to the desired outcome in a given situation." Bandura divided self-efficacy into two subcomponents, efficacy and outcome expectancy, and tried to explain human behaviour in this way. While efficacy expectancy describes the individual's belief that they can perform certain behaviours successfully (e.g., the woman's belief that she can successfully perform relaxation exercises during labour), outcome expectancy refers to the belief that performing a behaviour will lead to a result. (e.g., the woman's belief that she will experience less pain if she relaxes during labour). Self-efficacy is important in determining the direction of emotions, thoughts and behaviour patterns. For this reason, the "concept of birth self-efficacy" has been defined separately. Childbirth self-efficacy refers to the woman's self-confidence in coping with labour. Women with higher self-efficacy expectations are more likely to initiate and maintain pain-coping strategies. High childbirth self-efficacy is associated with improved perinatal outcomes and maternal health. A woman's self-confidence increases her access to methods of coping with labour and her ability to cope with the fear of birth. For this reason, it is important to associate the resources that nourish the concept of self-efficacy with childbirth. For this reason, Lowe associated self-efficacy resources with childbirth.Prenatal education is accepted as an effective strategy to improve women's self-efficacy during pregnancy. Prenatal education enables expectant mothers to make safe decisions during pregnancy and birth, improves their skills in coping with labour pain, increases birth self-efficacy and reduces the fear of birth. There are also study results showing that prenatal education can affect the type of birth, the use of birth-related interventions, and obstetric outcomes. It is especially important in terms of reducing the rate of interventional childbirth and cesarean sections. In recent years, yoga has been one of the preferred practices in the prenatal period due to its positive physical and psychological effects. Women see yoga as a holistic practice that can meet their needs during pregnancy, birth and the postpartum period. Despite the physiological effects of breathing exercises and yoga postures on the body during yoga practice, studies are often interested in the psychological effects of yoga. However, study results show that yoga performed during pregnancy can reduce pregnancy-related physiological disorders, shorten childbirth times, reduce childbirth pain, and increase childbirth self-efficacy and vaginal birth rate. Yoga provides somatic body awareness, especially with the meditation and breathing exercises it includes. Awareness of the body's physiological and psychological changes increases women's self-efficacy during childbirth. Considering this aspect, there are gaps in the literature regarding the effect of yoga during pregnancy on women's self

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous
* Being between the ages of 18 -35
* Having a single and healthy fetus
* 24-32. being in the pregnancy week
* Being no psychiatric diagnosis or treatment
* Using an online meeting program (Zoom®)

Exclusion Criteria:

* Women doing body-mind-based exercises (yoga, meditation, progressive muscle relaxation, mindfulness, etc.).
* Women taking birth preparation training
* Women having a regular exercise habit of approximately 90-150 minutes per week
* Women with a high-risk pregnancy diagnosis
* Having become pregnant through assisted reproductive techniques
* According to the Wijma delivery expectancy questionnaire-A scale score, women with severe fear of childbirth will be excluded and referred to psychiatry.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between the ages of 18-35 and have a single and healthy fetus at 24-32 weeks of gestation will be included in the study.
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Fear of Childbirth | Measurements will be taken at registration when participants are included in the study, and 6 weeks after the first measurement
  Fear of Childbirth (Measurement will be made using the Wijma Birth Expectation/Experience Scale A version. In the 6-point Likert type scale, 0 means "completely", and 5 means "not at all". The lowest score that can be obtained from the scale is 0, while the highest score is 165. It is interpreted that as the score obtained from the scale increases, the fear of birth experienced by women increases.)
Childbirth Self Efficacy | Measurements will be taken at registration when participants are included in the study, and 6 weeks after the first measurement
  Childbirth self-efficacy (Measurements will be made with the Childbirth Self Efficacy Scale-Short Form. The scale has two sub-dimensions. Each item is scored between 1 and 10 on the Likert-type scale. The lowest score on the scale is 32, and the highest If it is high, it is 320 points. As the total score obtained from the scale increases, self-efficacy regarding birth increases.)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İ̇zmi̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to roll out IPD.